CLINICAL TRIAL: NCT04324281
Title: Double Crush Syndrome in Median Nerve-cadaveric Observational Study
Brief Title: Myth of Double Crush Syndrome in Median Nerve
Acronym: cadaveric
Status: Completed | Type: Observational
Sponsor: Sahar Ahmed Abdalbary (Other)
Responsible Party: Sponsor-Investigator, Sahar Ahmed Abdalbary, Associate professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Cadaveric
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cervical Radiculopathy; Median Nerve Disease
Keywords: Wrist Pain
MeSH Terms: conditions — Radiculopathy; Median Neuropathy | interventions — Contact Tracing; Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Investigation — cadaveric dissection
  Other Names: observation

SUMMARY:
There is relation between the cervical radiculopathy and carpal tunnel syndrome and why the referred pain is fall at carpal tunnel not at elbow.

DETAILED DESCRIPTION:
This is an observational cadaveric study which examined median nerve from shoulder to wrist by histological measurements to explain the difference at the median nerve.

ELIGIBILITY:
Inclusion Criteria:

* Intact Upper Limb

Exclusion Criteria:

Amputation at upper limb

-

Ages: 35 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: They are people who wrote consent form before death to use there cadavers in medical research.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
histological study | 3 month
  Studying the histological structure of the median nerve at shoulder, elbow and wrist

CONTACTS AND LOCATIONS:
Locations (1):
- Sahar, Maadi, Egypt